CLINICAL TRIAL: NCT00407485
Title: A Phase II Study of VEGF Trap (NSC 724770) in Patients With Recurrent or Metastatic Transitional Carcinoma of the Urothelium
Brief Title: VEGF Trap in Treating Patients With Recurrent, Locally Advanced, or Metastatic Cancer of the Urothelium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02840; NCI-2012-02840 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHII-76 (Other: City of Hope); 7533 (Other: CTEP); N01CM62201 (NIH); N01CM62209 (NIH)
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Results first posted 2014-10-03 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2013-10

CONDITIONS: Adenocarcinoma of the Bladder; Distal Urethral Cancer; Metastatic Transitional Cell Cancer of the Renal Pelvis and Ureter; Proximal Urethral Cancer; Recurrent Bladder Cancer; Recurrent Transitional Cell Cancer of the Renal Pelvis and Ureter; Recurrent Urethral Cancer; Squamous Cell Carcinoma of the Bladder; Stage III Bladder Cancer; Stage III Urethral Cancer; Stage IV Bladder Cancer; Transitional Cell Carcinoma of the Bladder; Urethral Cancer Associated With Invasive Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — aflibercept

ARMS (1):
- Treatment (ziv-aflibercept) (Experimental): Patients receive 4 mg/kg VEGF Trap IV over 1 hour on day 1. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: ziv-aflibercept; Other: pharmacological study

INTERVENTIONS:
Biological: ziv-aflibercept — Given IV
Other: pharmacological study — Correlative studies

SUMMARY:
This phase II trial is studying the side effects and how well VEGF Trap works in treating patients with recurrent, locally advanced, or metastatic cancer of the urothelium. VEGF Trap may stop the growth of tumor cells by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate in patients with recurrent, locoregionally advanced, or metastatic transitional cell carcinoma of the urothelium treated with VEGF Trap.

II. Determine the time to progression in patients treated with this drug. III. Determine overall survival of patients treated with this drug. IV. Determine the tolerability and safety of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive VEGF Trap IV over 1 hour on day 1. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.

Patients undergo blood collection periodically during study for pharmacokinetic/pharmacodynamic correlative studies.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed transitional cell carcinoma (TCC) of the urothelium

  * Must have predominance of transitional histology, but foci of squamous and/or adenocarcinoma histology allowed
  * Poorly differentiated transitional cell carcinoma allowed
* TCC of any of the following sites allowed:

  * Bladder
  * Renal pelvis
  * Ureter
  * Urethra
* Measurable disease, defined as >= 1 unidimensionally measurable lesion >= 20 mm by conventional techniques OR >= 10 mm by spiral CT scan
* Locoregionally advanced or metastatic disease that is not amenable to curative surgery and/or radiotherapy
* Must have received 1 prior systemic chemotherapy regimen containing a platinum compound (e.g., cisplatin, carboplatin, or oxaliplatin) in the neoadjuvant, adjuvant, or metastatic setting
* No evidence of CNS disease, including primary brain tumor or brain metastases
* ECOG performance status 0-2
* Absolute neutrophil count >= 1,000/mm^3
* Platelet count >= 75,000/mm^3
* Bilirubin =< 1.5 times upper limit of normal (ULN)
* AST or ALT =< 2.5 times ULN
* Creatinine =< 2.5 times ULN OR creatinine clearance => 40 mL/min
* Urine protein: creatinine ratio =< 1 OR 24-hour urine protein < 500 mg
* INR =< 1.5 (unless on full-dose warfarin)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for >= 6 months after completion of study treatment
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to other agents used in the study
* No serious or nonhealing wound, ulcer, or bone fracture
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
* No significant traumatic injury within the past 28 days
* No clinically significant cardiovascular disease, including any of the following:

  * Myocardial infarction, coronary artery bypass graft, or unstable angina pectoris within the past 6 months
  * New York Heart Association class III or IV congestive heart failure
  * Serious cardiac arrhythmia requiring medication
  * Clinically significant peripheral vascular disease within the past 6 months
  * Cerebrovascular accident within the past 6 months
  * Pulmonary embolism, deep vein thrombosis, or other thromboembolic event within the past 6 months
  * Uncontrolled hypertension, defined as blood pressure (BP) > 150/100 mm Hg or systolic BP > 180 mm Hg (if diastolic BP < 90 mm Hg) within the past 3 months
* No evidence of bleeding diathesis or coagulopathy
* No uncontrolled intercurrent illness, including, but not limited to, any of the following:

  * Ongoing or active infection
  * Psychiatric illness or social situation that would preclude study compliance
* Recovered from prior therapy
* Prior biologic or targeted therapies allowed
* No more than 1 prior systemic chemotherapy regimen for metastatic disease
* No prior antiangiogenic therapy primarily targeting the vascular endothelial growth factor pathway
* At least 4 weeks since prior radiotherapy or systemic therapy (6 weeks for mitomycin C or nitrosoureas)
* More than 28 days since prior major surgery or open biopsy
* More than 7 days since prior core biopsy
* No concurrent major surgery
* Concurrent full-dose anticoagulants (e.g., warfarin) allowed provided all of the following criteria are met:

  * In-range INR (usually between 2 and 3) on a stable dose of oral anticoagulant or low molecular weight heparin
  * No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-11; Primary Completion 2010-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Przemyslaw Twardowski, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Ziv-aflibercept)
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ziv-aflibercept)
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 67 [45 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 15
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 20
  Americian Indian | 1
  Pacific Islander | 1
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate
Description: Response rate (RR) and progression free survival (PFS) were assessed in a 2-stage accrual design (22+18). A maximum of 40 patients were to be accrued to rule out a null hypothesized RR of 4% and PFS of 3 months versus alternative of 15% RR and 5.4 months PFS (corresponding to 4 month PFS of 40% vs 60%) with α=0.12 and β=0.19. If no more than 1 objective response (no more than 4.5%), and no more than 10 instances of 4-month PFS (no more than 45%), were observed among the initial 22 patients, the study would be terminated early and declared negative. Tumor response was evaluated by CT or MRI using RECIST v1.0 criteria.
  Responders were confirmed partial or complete responses to treatment.
Time Frame: From the start of the treatment until disease progression or recurrence, assessed up to 4 years
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Treatment (Ziv-aflibercept)
Number analyzed (Participants) | 22
percentage of responders | 4.5 [0.1 to 22.8]

2. Primary Outcome: Progression-free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions PFS using the product-limit method of Kaplan and Meier.
Time Frame: From start of treatment to time of progression, assessed up to 4 months
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Treatment (Ziv-aflibercept): Patients receive VEGF Trap IV over 1 hour on day 1. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.
  ziv-aflibercept: Given IV
  pharmacological study: Correlative studies
Arm/Group | Treatment (Ziv-aflibercept)
Number analyzed (Participants) | 22
Months | 2.79 [1.74 to 3.88]

ADVERSE EVENTS:
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Treatment (Ziv-aflibercept)
Serious Adverse Events (participants affected / at risk) | 4/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ziv-aflibercept) (N=22)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ziv-aflibercept) (N=22)
Hemoglobin decreased (Blood and lymphatic system disorders) | 12 (34)
Abdominal pain (Gastrointestinal disorders) | 3 (5)
Constipation (Gastrointestinal disorders) | 7 (11)
Diarrhea (Gastrointestinal disorders) | 6 (13)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (3)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (4)
Nausea (Gastrointestinal disorders) | 8 (10)
Oral pain (Gastrointestinal disorders) | 2 (2)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5)
Chills (General disorders) | 2 (3)
Death (General disorders) | 7 (7)
Disease progression (General disorders) | 2 (2)
Edema limbs (General disorders) | 2 (4)
Fatigue (General disorders) | 16 (51)
Pain (General disorders) | 3 (7)
Bladder infection (Infections and infestations) | 1 (2)
Sinusitis (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 9 (21)
Alkaline phosphatase increased (Investigations) | 8 (31)
Aspartate aminotransferase increased (Investigations) | 9 (16)
Bilirubin increased (Investigations) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 13 (42)
Leukocyte count decreased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 8 (21)
Platelet count decreased (Investigations) | 1 (4)
Weight loss (Investigations) | 3 (5)
Anorexia (Metabolism and nutrition disorders) | 10 (29)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 2 (4)
Blood glucose increased (Metabolism and nutrition disorders) | 14 (34)
Blood uric acid increased (Metabolism and nutrition disorders) | 3 (9)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 7 (13)
Serum calcium decreased (Metabolism and nutrition disorders) | 5 (10)
Serum calcium increased (Metabolism and nutrition disorders) | 2 (2)
Serum glucose decreased (Metabolism and nutrition disorders) | 4 (4)
Serum phosphate decreased (Metabolism and nutrition disorders) | 5 (7)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (3)
Serum potassium increased (Metabolism and nutrition disorders) | 8 (15)
Serum sodium decreased (Metabolism and nutrition disorders) | 8 (15)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (18)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 4 (9)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (7)
Dizziness (Nervous system disorders) | 3 (4)
Headache (Nervous system disorders) | 10 (20)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (4)
Taste alteration (Nervous system disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Hemoglobin urine positive (Renal and urinary disorders) | 1 (2)
Hemorrhage urinary tract (Renal and urinary disorders) | 5 (9)
Protein urine positive (Renal and urinary disorders) | 8 (17)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 4 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (4)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (3)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (3)
Hypertension (Vascular disorders) | 14 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less